CLINICAL TRIAL: NCT01621802
Title: Immunogenicity and Safety Study of GSK Biologicals' Combined Measles-mumps-rubella Vaccine in Subjects Four to Six Years of Age (209762)
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Combined Measles-mumps-rubella (MMR) Vaccine in Subjects Four to Six Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115158; 2011-004638-32 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Measles-Mumps-Rubella
Keywords: Safety; Measles, mumps and rubella diseases; Immunogenicity
MeSH Terms: conditions — Measles; Mumps | interventions — Measles-Mumps-Rubella Vaccine; DTPP vaccine; measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Inv _MMR_CO Group (Experimental): Subjects received one dose of the study vaccine Priorix along with Kinrix and ProQuad vaccines at Visit 1 (Day 0).
  Interventions: Biological: Priorix; Biological: Kinrix; Biological: ProQuad
- Com_MMR_CO Group (Active Comparator): Subjects received one dose of the licensed vaccine M-M-R II (also known as M-M-R Vax Pro) Lot 1 or Lot 2 along with Kinrix and ProQuad vaccines at Visit 1 (Day 0).
  Interventions: Biological: M-M-R II; Biological: Kinrix; Biological: ProQuad
- Inv_MMR_I Group (Experimental): Subjects received one dose of Priorix at Visit 1 (Day 0).
  Interventions: Biological: Priorix
- Com_MMR_I Group (Active Comparator): Subjects received one dose of M-M-R II (also known as M-M-R Vax Pro) vaccine from Lot 1 or Lot 2 at Visit 1 (Day 0).
  Interventions: Biological: M-M-R II
- Inv _MMR_S Group (Experimental): Subjects in this safety cohort received one dose of Priorix at Visit 1 (Day 0).
  Interventions: Biological: Priorix
- Com_MMR_S Group (Active Comparator): Subjects in this safety cohort received one dose of M-M-R II (also known as M-M-R Vax Pro) vaccine from Lot 1 or Lot 2 at Visit 1 (Day 0).
  Interventions: Biological: M-M-R II

INTERVENTIONS:
Biological: Priorix — One dose administered subcutaneously in the triceps region of the right arm.
  Arms: Inv _MMR_CO Group; Inv _MMR_S Group; Inv_MMR_I Group
Biological: M-M-R II — One dose administered subcutaneously in the triceps region of the right arm.
  Arms: Com_MMR_CO Group; Com_MMR_I Group; Com_MMR_S Group
Biological: Kinrix — One dose administered by deep intramuscular injection in the upper left deltoid.
  Arms: Com_MMR_CO Group; Inv _MMR_CO Group
Biological: ProQuad — One dose administered subcutaneously in the triceps region of the left arm.
  Arms: Com_MMR_CO Group; Inv _MMR_CO Group

SUMMARY:
The purpose of this study is to support licensure of GSK Biologicals' MMR vaccine (Priorix®) in the US by generating immunogenicity and safety data in contrast to the US standard of care, Merck's MMR vaccine (M-M-R®II), when given as a second dose to children four to six years of age.

DETAILED DESCRIPTION:
The GSK Biologicals' MMR vaccine (Priorix®) and Merck's MMR vaccine (M-M-R®II) are referred to as Inv_MMR vaccine and Com_MMR vaccine respectively. 2 lots of the comparator vaccine (Com_MMR_L1 and Com_MMR_L2) will be used, but the 2 lots will be analysed as a pool.

The Inv_MMR vaccine will be administered as a second dose to children who already received a first dose Com_MMR vaccine. Since the second dose of a MMR vaccine in the US is routinely co-administered with DTaP-IPV vaccine (Kinrix®) and varicella vaccine (VV) (ProQuad® or Varivax®), some children will receive one dose of these vaccines along with either of the MMR vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s) or LAR/s can and will comply with the requirements of the protocol.
* Male or female subjects 4 to 6 years of age at the time of vaccination.
* Written informed consent is obtained from the parent(s)/LAR(s) of the subject (assent will be obtained from subjects in line with local rules and regulations).
* Subjects in stable health as determined by investigator's physical examination and assessment of subjects' medical history.
* Subjects received either a single dose of M-M-R II, M-M-R VaxPro or ProQuad in the second year of life.
* For subjects enrolled in the sub-cohort receiving co-administered DTaP-IPV and VV:

  * subjects received previous DTaP vaccine doses with INFANRIX® and/or PEDIARIX® for the first three doses and INFANRIX® for the fourth dose of the DTaP-containing vaccine.
  * subjects received a first dose of VV in the second year of life.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the day of study vaccination/s or planned during the entire study period.
* Previous vaccination with a second dose of measles, mumps, rubella containing vaccine/s.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to Day 0 or any planned administration of immunosuppressive and immune-modifying drugs during the entire study. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products during the period starting 180 days before entering the study or planned administration from the date of vaccination through the immunogenicity evaluation at Visit 2.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days prior to the study vaccination/s and ending 42 days after the vaccination/s (at Visit 2), with the exception of live intranasal or inactivated influenza (flu) vaccine, which may be given at any time during the study, including the day of study vaccination/s. Inactivated influenza vaccine must be administered at a different location from the study vaccine. Any age appropriate vaccine may be given starting at Visit 2, and anytime thereafter.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of measles, mumps, and/or rubella disease.
* Known exposure to measles, mumps and/or rubella during the period starting 30 days prior to enrollment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including systemic hypersensitivity to neomycin or gelatin.
* Blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Fever is defined as temperature ≥38°C (100.4°F) measured by any age appropriate route. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection without fever.
* Active untreated tuberculosis according to the subject's medical history.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

In addition, for subjects enrolled in the sub-cohort receiving co-administered DTaP-IPV+VV:

* Previous vaccination with a second dose of varicella-containing vaccine.
* Receipt of any varicella-containing vaccine during the period starting 90 days before the day of study vaccination.
* History of varicella/zoster disease.
* Known exposure to varicella/zoster during the period starting 30 days prior to enrollment.
* History of diphtheria, tetanus, pertussis, and/or poliomyelitis disease.
* Vaccination against diphtheria, tetanus, pertussis or polio given after the second year of life.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunization against diphtheria and/or tetanus toxoids.
* Following a previous administration of DTP vaccine: temperature ≥40.6°C (>105°F) during the period starting 48 hours not due to another identifiable cause, collapse or shock-like state during the period starting 48 hours, persistent, inconsolable crying lasting three hours or more within 48 hours, seizures with or without fever occurring during the period starting three days, or encephalopathy of unknown aetiology occurring during the period starting 7 days of a previous administration of DTP vaccine.
* Hypersensitivity reaction to any component of the DTaP-IPV and/or varicella vaccines.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4011 (Actual)
Dates: Start 2012-06-21 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (60):
- United States (47):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Baldwin Park, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Augusta, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Cheraw, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Monroe, Wisconsin
- South Korea (9):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, GyeongSangNam-do
  - GSK Investigational Site, Iksan
  - GSK Investigational Site, Jeollabukdo
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wonju-si Kangwon-do
- Taiwan (4):
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19838

REFERENCES:
- [Background] MMR-158 Study Group. A second dose of a measles-mumps-rubella vaccine administered to healthy four-to-six-year-old children: a phase III, observer-blind, randomized, safety and immunogenicity study comparing GSK MMR and MMR II with and without DTaP-IPV and varicella vaccines co-administration. Hum Vaccin Immunother. 2019;15(4):786-799. doi: 10.1080/21645515.2018.1554971. Epub 2019 Feb 20. PMID 30785357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in 3 sub-cohorts. Sub-cohort 1: Inv_MMR_CO and Com_MMR_CO (Lot 1 or Lot 2), Sub-cohort 2: Inv_MMR_I and Com_MMR_I (Lot 1 or Lot 2) and Sub-cohort 3: Inv_MMR_S and Com_MMR_S (Lot 1 or Lot 2).
Pre-assignment Details: 4011 subjects were enrolled in the study with 4007 eligible subjects receiving a study vaccination.
Groups:
- Inv_MMR_CO Group: Subjects received one dose of the study vaccine Priorix along with Kinrix and ProQuad vaccines at Visit 1 (Day 0).
- Inv_MMR_S Group: Subjects in this safety cohort received one dose of Priorix at Visit 1 (Day 0).
Period: Overall Study
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Started | 802 | 298 | 796 | 303 | 1319 | 489
Completed | 755 | 275 | 763 | 292 | 1284 | 477
Not Completed | 47 | 23 | 33 | 11 | 35 | 12
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 4 | 4 | 2 | 2 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Others | 3 | 3 | 3 | 2 | 1 | 0
Not completed — Lost to Follow-up | 36 | 16 | 24 | 7 | 31 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group | Total
Number analyzed (Participants) | 802 | 298 | 796 | 303 | 1319 | 489 | 4007
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.1 (0.3) | 4.1 (0.3) | 4.4 (0.6) | 4.3 (0.6) | 4.4 (0.6) | 4.4 (0.6) | 4.3 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398 | 134 | 361 | 153 | 632 | 225 | 1903
  Male | 404 | 164 | 435 | 150 | 687 | 264 | 2104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African Heritage / African American | 96 | 39 | 48 | 19 | 94 | 32 | 328
  Race/Ethnicity: American Indian or Alaskan Native | 130 | 38 | 15 | 3 | 4 | 0 | 190
  Race/Ethnicity: Asian - Central/South Asian Heritage | 12 | 5 | 7 | 1 | 8 | 0 | 33
  Race/Ethnicity: Asian - East Asian Heritage | 28 | 6 | 384 | 146 | 565 | 209 | 1338
  Race/Ethnicity: Asian - Japanese Heritage | 3 | 0 | 0 | 1 | 1 | 0 | 5
  Race/Ethnicity: Asian - South East Asian Heritage | 49 | 25 | 11 | 4 | 16 | 8 | 113
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 4 | 2 | 2 | 0 | 3 | 0 | 11
  Race/Ethnicity: Other | 112 | 45 | 35 | 9 | 52 | 22 | 275
  Race/Ethnicity: White - Arabic / North African Heritage | 5 | 3 | 3 | 3 | 1 | 0 | 15
  Race/Ethnicity: White - Caucasian / European Heritage | 363 | 135 | 291 | 117 | 575 | 218 | 1699

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-measles virus antibody concentration equal to or above (≥) 200 milli-international Units per milliliter (mIU/mL). Analysis was done in sub-cohorts 1 and 2 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: This analysis was performed on According to Protocol (ATP) cohort for immunogenicity which included all evaluable subjects with post-vaccination serology results available for measles vaccine component, did not meet any elimination criteria up to Visit 2 blood sample & complied with protocol procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group
Number analyzed (Participants) | 697 | 249 | 736 | 283
Participants | 697 | 249 | 736 | 281
Statistical Analysis 1: Comparison: Inv_MMR_CO Group vs Com_MMR_CO Group; Power obtained using PASS 2005 (Likelihood Score [Miettienen and Nurminen approach]), one-sided non-inferiority test for the difference of two independent proportions, under the alternative associated to the reference value & alpha=1.25%. The global power to reach all non-inferiority objectives of Priorix vs. M-M-R II in sub-cohort 1 should be at least 94.04% (=100%- the sum of type II errors associated to cohort 1; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion for sub cohort 1: Lower limit (LL) of the 2-sided 97.5% confidence interval (CI) for group difference (Inv_MMR_CO Group minus pooled Com_MMR_CO Group) in seroresponse rates to measles, mumps and rubella viruses is ≥ -5%; Difference in seroresponse rate (%) = 0.00, 97.5% CI 2-sided [-0.72 to 1.98] — Difference in percentage (Inv_MMR_CO Group minus Com_MMR_CO Group) in percentage of subjects with an anti-measles antibody concentration ≥ 200 mIU/mL
Statistical Analysis 2: Comparison: Inv_MMR_I Group vs Com_MMR_I Group; Power obtained using PASS 2005 (Likelihood Score [Miettienen and Nurminen approach]), one-sided non-inferiority test for the difference of two independent proportions, under the alternative associated to the reference value & alpha=1.25%. The global power to reach all non-inferiority objectives of Priorix vs. M-M-R II in sub-cohort 2 should be at least 98.88% (=100%- the sum of type II error associated to cohort 2; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion for sub cohort 2: The LL of the 2-sided 97.5% CI for group difference (Inv_MMR_I group minus pooled Com_MMR_I group) in seroresponse rates to measles, mumps and rubella viruses was ≥ -5%; Difference in Seroresponse rate (%) = 0.71, 97.5% CI 2-sided [0.02 to 2.97] — Difference in percentage (Inv_MMR_I Group minus Com_MMR_I Group) in percentage of subjects with an anti-Measles antibody concentration ≥ 200 mIU/mL

2. Primary Outcome: Number of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥ 10 ELISA Units per milliliter (EU/mL). Analysis was done in sub-cohorts 1 and 2 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: This analysis was performed on ATP cohort for immunogenicity which included all evaluable subjects with post-vaccination serology results available for mumps vaccine component, did not meet any elimination criteria up to Visit 2 blood sample & complied with protocol procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group
Number analyzed (Participants) | 698 | 250 | 736 | 283
Participants | 698 | 250 | 736 | 283
Statistical Analysis 1: Comparison: Inv_MMR_CO Group vs Com_MMR_CO Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion for sub cohort 1: The LL of the 2-sided 97.5% CI for group difference (Inv_MMR_CO Group minus pooled Com_MMR_CO Group) in seroresponse rates to measles, mumps and rubella viruses was ≥ -5%; Difference in seroresponse rate (%) = 0.00, 97.5% CI 2-sided [-0.72 to 1.97] — Difference in percentage (Inv_MMR_CO Group minus Com_MMR_CO Group) in percentage of subjects with an anti-mumps antibody concentration ≥ 10 EU/mL
Statistical Analysis 2: Comparison: Inv_MMR_I Group vs Com_MMR_I Group; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference in Seroresponse rate (%) = 0.00, 97.5% CI 2-sided [-0.68 to 1.75] — Difference in percentage (Inv_MMR_I Group minus Com_MMR_I Group) in percentage of subjects with an anti-mumps antibody concentration ≥ 10 EU/mL

3. Primary Outcome: Number of Subjects With Anti-rubella Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-rubella virus antibody concentration ≥ 10 International Units per milliliter (IU/mL). Analysis was done in sub-cohorts 1 and 2 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: This analysis was performed on ATP cohort for immunogenicity which included all evaluable subjects with post-vaccination serology results available for rubella vaccine component, did not meet any elimination criteria up to Visit 2 blood sample & complied with protocol procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group
Number analyzed (Participants) | 697 | 249 | 736 | 283
Participants | 696 | 249 | 736 | 283
Statistical Analysis 1: Comparison: Inv_MMR_CO Group vs Com_MMR_CO Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in seroresponse rate (%) = -0.14, 97.5% CI 2-sided [-0.98 to 1.84] — Difference in percentage (Inv_MMR_CO Group minus Com_MMR_CO Group) in percentage of subjects with an anti-rubella antibody concentration ≥ 10 IU/mL
Statistical Analysis 2: Comparison: Inv_MMR_I Group vs Com_MMR_I Group; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference in seroresponse rate (%) = 0.00, 97.5% CI 2-sided [-0.68 to 1.75] — Difference in percentage (Inv_MMR_I Group minus Com_MMR_I Group) in percentage of subjects with an anti-rubella antibody concentration ≥ 10 IU/mL

4. Primary Outcome: Evaluation of Immunogenicity in Terms of Anti-measles Virus Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. Analysis was done in sub-cohorts 1 and 2 only.
Time Frame: 42 days after vaccination (At Day 42)
Population: This analysis was performed on ATP cohort for immunogenicity which included all evaluable subjects with post-vaccination serology results available for measles vaccine component, did not meet any elimination criteria up to Visit 2 blood sample & complied with protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group
Number analyzed (Participants) | 697 | 249 | 736 | 283
mIU/mL | 4335.0 [4089.7 to 4594.9] | 4215.6 [3806.7 to 4668.4] | 3646.6 [3453.5 to 3850.4] | 3503.9 [3174.6 to 3867.4]
Statistical Analysis 1: Comparison: Inv_MMR_CO Group vs Com_MMR_CO Group; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion for sub cohort 1: The LL of the 2-sided 97.5% CI for the adjusted GMC ratio (Inv_MMR_CO group divided by pooled Com_MMR_CO group) was ≥ 0.67 for antibodies to measles, mumps and rubella viruses; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 0.99, 97.5% CI 2-sided [0.92 to 1.06] — The GMCs were used to calculate the Adjusted GMCs, which in turn were used to calculate the Adjusted GMC ratio with 97.5% confidence interval
Statistical Analysis 2: Comparison: Inv_MMR_I Group vs Com_MMR_I Group; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion for sub cohort 2: The LL of the 2-sided 97.5% CI for the adjusted GMC ratio (Inv_MMR_I group divided by pooled Com_MMR_I group) was ≥ 0.67 for antibodies to measles, mumps and rubella viruses; ANCOVA; Ancova model: adjustment for baseline concentration country - pooled variance; Adjusted GMC ratio = 1.03, 97.5% CI 2-sided [0.96 to 1.10] — [estimate comment as in outcome 4, analysis 1]

5. Primary Outcome: Evaluation of Immunogenicity in Terms of Anti-mumps Virus Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in EU/mL. Analysis was done in sub-cohorts 1 and 2 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group
Number analyzed (Participants) | 698 | 250 | 736 | 283
EU/mL | 170.5 [161.6 to 179.9] | 190.1 [174.7 to 206.8] | 167.2 [158.6 to 176.3] | 176.2 [161.5 to 192.2]
Statistical Analysis 1: Comparison: Inv_MMR_CO Group vs Com_MMR_CO Group; Test type: Non-Inferiority or Equivalence — The LL of the 2-sided 97.5% CI for the adjusted GMC ratio (Inv_MMR_CO group divided by pooled Com_MMR_CO group) was ≥ 0.67 for antibodies to measles, mumps and rubella viruses; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 0.91, 97.5% CI 2-sided [0.83 to 1.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Inv_MMR_I Group vs Com_MMR_I Group; Test type: Non-Inferiority or Equivalence — The LL of the 2-sided 97.5% CI for the adjusted GMC ratio (Inv_MMR_I group divided by pooled Com_MMR_I group) was ≥ 0.67 for antibodies to measles, mumps and rubella viruses; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 0.96, 97.5% CI 2-sided [0.87 to 1.06] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: Evaluation of Immunogenicity in Terms of Anti-rubella Virus Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in IU/mL. Analysis was done in sub-cohorts 1 and 2 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group
Number analyzed (Participants) | 697 | 249 | 736 | 283
IU/mL | 96.4 [92.6 to 100.4] | 96.0 [89.5 to 103.0] | 98.9 [95.3 to 102.8] | 98.7 [93.2 to 104.5]
Statistical Analysis 1: Comparison: Inv_MMR_CO Group vs Com_MMR_CO Group; Adjusted geometric mean concentration (GMC) ratio (Inv_MMR_CO group divided by Com_MMR_CO group) for antibodies to rubella virus; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 1.03, 97.5% CI 2-sided [0.97 to 1.09] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Inv_MMR_I Group vs Com_MMR_I Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 2]; ANCOVA; Ancova model: adjustment for baseline concentration - pooled variance; Adjusted GMC ratio = 1.01, 97.5% CI 2-sided [0.95 to 1.07] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Number of Subjects With Anti-varicella Zoster Virus (VZV) Antibody Concentration Equal to or Above the Cut-off-value
Description: Seroresponse was defined as post-vaccination anti-VZV antibody concentration ≥ 75 mIU/mL. Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: This analysis was performed on ATP cohort for immunogenicity which included all evaluable subjects with post-vaccination serology results available for at least one of the three vaccine components (measles, mumps, or rubella), did not meet any elimination criteria up to Visit 2 blood sample & complied with protocol procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 695 | 247
Participants | 693 | 247

8. Secondary Outcome: Evaluation of Immunogenicity in Terms of Anti-VZV Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in mIU/mL. Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 695 | 247
mIU/mL | 887.7 [834.3 to 944.4] | 820.4 [749.3 to 898.3]

9. Secondary Outcome: Number of Subjects With Antibody Booster Response to Diphtheria Toxin (Anti-D) and Tetanus Toxin (Anti-T)
Description: Booster response was defined as:
  For subjects with pre-vaccination antibody concentration less than (<) 0.1 IU/mL, antibody concentration ≥ 0.4 IU/ml at Day 42.
  For subjects with pre-vaccination antibody concentration ≥ 0.1 IU/mL: antibody concentration at Day 42 ≥ 4 fold the pre-vaccination antibody concentration.
  Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 661 | 234
Participants
  Anti-D: number analyzed (Participants) | 659 | 233
  Anti-D | 657 | 233
  Anti-T | 621 | 224

10. Secondary Outcome: Number of Subjects With Antibody Booster Response to Pertussis Toxin (PT)
Description: Booster response was defined as:
  For initially seronegative subjects, antibody concentration ≥ 10.772 IU/mL at Day 42.
  For initially seropositive subjects with pre-vaccination antibody concentration < 10.772 IU/mL: antibody concentration at Day 42 ≥ 4 fold the pre-vaccination antibody concentration.
  For initially seropositive subjects with pre-vaccination antibody concentration ≥ 10.772 IU/mL: antibody concentration at Day 42 ≥ 2 fold the pre-vaccination antibody concentration.
  Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 659 | 233
Participants | 643 | 225

11. Secondary Outcome: Number of Subjects With Antibody Booster Response to Filamentous Hemagglutinin (FHA)
Description: Booster response was defined as:
  For initially seronegative subjects, antibody concentration ≥ 8.184 IU/ml at Day 42.
  For initially seropositive subjects with pre-vaccination antibody concentration < 8.184 IU/mL: antibody concentration at Day 42 ≥ 4 fold the pre-vaccination antibody concentration.
  For initially seropositive subjects with pre-vaccination antibody concentration ≥ 8.184 IU/mL: antibody concentration at Day 42 ≥ 2 fold the pre-vaccination antibody concentration.
  Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 659 | 234
Participants | 620 | 221

12. Secondary Outcome: Number of Subjects With Antibody Booster Response to Pertactin (PRN)
Description: Booster response was defined as:
  For initially seronegative subjects, antibody concentration ≥ 8.748 IU/mL at Day 42.
  For initially seropositive subjects with pre-vaccination antibody concentration < 8.748 IU/mL: antibody concentration at Day 42 ≥ 4 fold the pre-vaccination antibody concentration.
  For initially seropositive subjects with pre-vaccination antibody concentration ≥ 8.748 IU/mL: antibody concentration at Day 42 ≥ 2 fold the pre-vaccination antibody concentration.
  Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 660 | 234
Participants | 657 | 233

13. Secondary Outcome: Evaluation of Immunogenicity in Terms of Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in IU/mL. Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 684 | 243
IU/mL
  Anti-D | 17.2 [16.2 to 18.1] | 17.8 [16.1 to 19.6]
  Anti-T | 7.4 [6.9 to 7.8] | 8.4 [7.6 to 9.3]

14. Secondary Outcome: Evaluation of Immunogenicity in Terms of Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs in EU/mL. Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 684 | 243
EU/mL
  Anti-PT | 76.6 [71.6 to 82.0] | 73.9 [66.2 to 82.4]
  Anti-FHA | 316.2 [299.4 to 334.0] | 319.3 [293.1 to 347.9]
  Anti-PRN: number analyzed (Participants) | 682 | 243
  Anti-PRN | 402.2 [370.4 to 436.8] | 427.3 [377.6 to 483.4]

15. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations ≥ 0.1 IU/mL
Description: Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 684 | 243
Participants
  Anti-D | 684 | 243
  Anti-T | 684 | 243

16. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations ≥ 1.0 IU/mL
Description: Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 684 | 243
Participants
  Anti-D | 683 | 242
  Anti-T | 678 | 243

17. Secondary Outcome: Evaluation of Immunogenicity in Terms of Anti-polio Virus Types 1, 2 and 3 Antibody Titers
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs) in ED50. Analysis was done in sub-cohort 1 only.
Time Frame: 42 days post vaccination (At Day 42)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ED50
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 669 | 238
ED50
  Anti-Polio 1 | 1618.7 [1499.8 to 1747.0] | 1587.3 [1387.3 to 1816.1]
  Anti-Polio 2: number analyzed (Participants) | 653 | 233
  Anti-Polio 2 | 2026.4 [1881.2 to 2182.7] | 2206.1 [1955.2 to 2489.3]
  Anti-Polio 3: number analyzed (Participants) | 590 | 214
  Anti-Polio 3 | 2753.5 [2512.4 to 3017.6] | 3040.6 [2613.0 to 3538.1]

18. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 Pain = Cried when limb was moved/spontaneously painful. Grade 3 redness and swelling = greater than 50 millimeters (m m ) i.e . > 50mm.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: This analysis was performed on Total Vaccinated cohort which included all vaccinated subjects with at least one vaccine administration documented. Analysis of the solicited symptoms based on the Total Vaccinated cohort included only subjects/doses with documented safety data (i.e., symptom screen/sheet completed).
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 727 | 267 | 766 | 289 | 1289 | 480
Participants
  Any Pain | 295 | 109 | 152 | 64 | 278 | 123
  Grade 3 Pain | 22 | 4 | 6 | 2 | 5 | 2
  Any Redness | 157 | 69 | 146 | 53 | 242 | 90
  Grade 3 Redness | 9 | 4 | 0 | 0 | 0 | 0
  Any Swelling | 82 | 28 | 64 | 23 | 108 | 42
  Grade 3 Swelling | 3 | 3 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 Drowsiness = Drowsiness that prevented normal activity, Grade 3 Loss of appetite = Not eating at all. Related = symptom assessed by the investigator as causally related to study vaccination.
  Analysis was done for sub-cohort 1 only.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group
Number analyzed (Participants) | 731 | 268
Participants
  Any Drowsiness | 199 | 72
  Grade 3 Drowsiness | 10 | 3
  Related Drowsiness | 180 | 63
  Any Loss of appetite | 154 | 59
  Grade 3 Loss of appetite | 2 | 2
  Related Loss of appetite | 135 | 56

20. Secondary Outcome: Number of Subjects Reporting Fever
Description: Any fever = fever ≥ 38°C; Grade 3 fever = fever > 39.5°C; Related = fever assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 731 | 268 | 767 | 291 | 1291 | 481
Participants
  Any fever | 177 | 67 | 146 | 58 | 257 | 96
  Grade 3 fever | 7 | 6 | 14 | 9 | 21 | 8
  Related fever | 100 | 32 | 27 | 11 | 52 | 25

21. Secondary Outcome: Number of Subjects Reporting MMR Specific Solicited General Symptoms
Description: Assessed MMR specific symptoms were parotid gland swelling and any suspected signs of meningism including febrile convulsions. Any = occurrence of any general symptoms regardless of their intensity grade or relationship to vaccination. Grade 3 Parotid/salivary gland swelling = Swelling accompanied with general symptoms. Grade 3 Sign of meningism (any suspected signs including febrile convulsions) = An event which prevented normal, everyday activities. Related = symptom assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 731 | 268 | 767 | 291 | 1291 | 481
Participants
  Any Sign of meningism | 0 | 2 | 1 | 0 | 0 | 0
  Grade 3 Sign of meningism | 0 | 0 | 0 | 0 | 0 | 0
  Related Sign of meningism | 0 | 2 | 0 | 0 | 0 | 0
  Any Parotid gland swelling | 0 | 0 | 0 | 1 | 1 | 1
  Grade 3 Parotid gland swelling | 0 | 0 | 0 | 0 | 0 | 0
  Related Parotid gland swelling | 0 | 0 | 0 | 1 | 1 | 1

22. Secondary Outcome: Number of Subjects Reporting Investigator-confirmed Rash
Description: Assessed any rash, varicella-like rash, measles/rubella-like rash, Grade 3, related. Any= occurrence of rash regardless of intensity grade. Grade 3 measles/rubella/varicella-like rash = Rash with more than 150 lesions. Other Grade 3 Rash = Rash that prevented normal, everyday activities. Related= Rash assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 731 | 268 | 767 | 291 | 1291 | 481
Participants
  Any localized or generalized | 61 | 28 | 37 | 12 | 56 | 23
  Any with fever | 11 | 7 | 5 | 1 | 6 | 1
  Any Varicella like | 4 | 3 | 0 | 0 | 0 | 0
  Any Measles/Rubella like | 14 | 5 | 3 | 2 | 4 | 2
  Any grade 3 | 3 | 0 | 1 | 0 | 3 | 0
  Any related | 25 | 11 | 2 | 2 | 8 | 3
  Localized any | 50 | 24 | 27 | 9 | 42 | 19
  Localized administration site | 9 | 2 | 1 | 0 | 8 | 0
  Localized other site | 41 | 22 | 26 | 9 | 36 | 19
  Localized with fever | 8 | 6 | 4 | 0 | 4 | 1
  Localized Varicella like | 2 | 2 | 0 | 0 | 0 | 0
  Localized Measles/Rubella like | 12 | 4 | 3 | 2 | 4 | 1
  Localized Grade 3 | 2 | 0 | 1 | 0 | 0 | 0
  Localized related | 18 | 10 | 2 | 2 | 7 | 2
  Generalized any | 12 | 4 | 10 | 3 | 15 | 4
  Generalized with fever | 3 | 1 | 1 | 1 | 2 | 0
  Generalized Varicella like | 2 | 1 | 0 | 0 | 0 | 0
  Generalized Measles/Rubella like | 2 | 1 | 0 | 0 | 0 | 1
  Generalized Grade 3 | 1 | 0 | 0 | 0 | 3 | 0
  Generalized Related | 7 | 1 | 0 | 0 | 1 | 1

23. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: During the entire study period (from Day 0 up to Day 180)
Population: This analysis was performed on Total Vaccinated cohort which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 802 | 298 | 796 | 303 | 1319 | 489
Participants | 8 | 4 | 6 | 0 | 11 | 3

24. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Description: The number of subjects reporting adverse events resulting in Emergency Room (ER) visits is reported.
Time Frame: During the entire study period (from Day 0 up to Day 180)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 802 | 298 | 796 | 303 | 1319 | 489
Participants | 61 | 29 | 64 | 22 | 102 | 36

25. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 802 | 298 | 796 | 303 | 1319 | 489
Participants | 276 | 90 | 314 | 112 | 508 | 186

26. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Any SAE = occurrence of SAE regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (from Day 0 up to Day 180)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Groups:
- Com_MMR_CO Group: Subjects received one dose of the licensed vaccine M-M-RII (also known as M-M-R Vax Pro) Lot 1 or Lot 2 along with Kinrix and ProQuad vaccines at Visit 1 (Day 0).
- Com_MMR_I Group: Subjects received one dose of M-M-RII (also known as M-M-R Vax Pro) vaccine from Lot 1 or Lot 2 at Visit 1 (Day 0).
- Com_MMR_S Group: Subjects in this safety cohort received one dose of M-M-RII (also known as M-M-R Vax Pro) vaccine from Lot 1 or Lot 2 at Visit 1 (Day 0).
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
Number analyzed (Participants) | 802 | 298 | 796 | 303 | 1319 | 489
Participants | 4 | 0 | 14 | 1 | 25 | 9

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms (drowsiness and loss of appetite): during the 4-day (Days 0-3) post-vaccination period; Solicited general and Unsolicited AEs: during the 43-day (Days 0-42) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Day 180).
Arm/Group | Inv_MMR_CO Group | Com_MMR_CO Group | Inv_MMR_I Group | Com_MMR_I Group | Inv_MMR_S Group | Com_MMR_S Group
All-Cause Mortality (participants affected / at risk) | 0/802 | 0/298 | 0/796 | 0/303 | 0/1319 | 0/489
Serious Adverse Events (participants affected / at risk) | 4/802 | 0/298 | 14/796 | 1/303 | 25/1319 | 9/489
Other Adverse Events (participants affected / at risk) | 544/802 | 198/298 | 410/796 | 156/303 | 702/1319 | 279/489
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inv_MMR_CO Group (N=802) | Com_MMR_CO Group (N=298) | Inv_MMR_I Group (N=796) | Com_MMR_I Group (N=303) | Inv_MMR_S Group (N=1319) | Com_MMR_S Group (N=489)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 5 (5) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (3)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inv_MMR_CO Group (N=802) | Com_MMR_CO Group (N=298) | Inv_MMR_I Group (N=796) | Com_MMR_I Group (N=303) | Inv_MMR_S Group (N=1319) | Com_MMR_S Group (N=489)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (41) | 16 (17) | 37 (41) | 8 (8) | 47 (50) | 21 (22)
Decreased appetite (Metabolism and nutrition disorders) | 156 (159) | 61 (61) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Injection site erythema (General disorders) | 170 (173) | 73 (75) | 147 (147) | 53 (53) | 242 (242) | 90 (90)
Injection site pain (General disorders) | 309 (321) | 118 (125) | 153 (153) | 64 (64) | 278 (278) | 123 (123)
Injection site swelling (General disorders) | 97 (97) | 31 (32) | 64 (64) | 23 (23) | 108 (108) | 42 (42)
Nasopharyngitis (Infections and infestations) | 25 (27) | 3 (3) | 77 (100) | 28 (32) | 112 (143) | 45 (57)
Pyrexia (General disorders) | 177 (177) | 67 (67) | 146 (146) | 58 (58) | 257 (257) | 96 (96)
Rash (Skin and subcutaneous tissue disorders) | 61 (61) | 28 (28) | 37 (37) | 12 (12) | 56 (56) | 23 (23)
Somnolence (Nervous system disorders) | 199 (199) | 73 (73) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 27 (28) | 11 (11) | 55 (66) | 27 (35) | 92 (107) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.